CLINICAL TRIAL: NCT06325813
Title: ADHD PreSMA Response Inhibition Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CIN001 - ADHD PreSMART
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active repetitive TMS (Active Comparator)
  Interventions: Device: Active repetitive TMS
- Sham repetitive TMS (Sham Comparator)
  Interventions: Device: Sham repetitive TMS

INTERVENTIONS:
Device: Active repetitive TMS — In this study, ADHD children will receive two trains of intermittent theta burst stimulation. Intermittent theta burst stimulation is a form of repetitive TMS. Both iTBS trains will be active stimulation using the active TMS coil.
  Arms: Active repetitive TMS
Device: Sham repetitive TMS — In this study, ADHD children will receive two trains of intermittent theta burst stimulation. Intermittent theta burst stimulation is a form of repetitive TMS. The first iTBS train will be sham stimulation using the sham TMS coil. The second iTBS train will be active stimulation using the active TMS coil.
  Arms: Sham repetitive TMS

SUMMARY:
ADHD children have abnormal inhibitory control, meaning they have trouble stopping themselves from doing something they should not do. This ability to control involves an area in the brain called the pre-supplementary motor area (pre-SMA). Scientists have previously shown that the pre-SMA is abnormal in ADHD patients. In this study, we will use Transcranial Magnetic Stimulation (TMS) to stimulate the pre-SMA and determine the effects on measures that are related to inhibitory control.

DETAILED DESCRIPTION:
ADHD children (ages 12-17 years) will be recruited. Cognitive testing and basic anatomic brain MRI will be performed during visit 1. During visit 2, baseline TMS-based physiologic measures will be obtained. Children will also complete a behavioral task (stop signal task) while electroencephalography (EEG) data is collected. After these baseline measures, two trains of Intermittent Theta Burst Stimulation (iTBS) will be delivered. (Intermittent Theta Burst Stimulation is a form of repetitive TMS.) The first train of iTBS will be randomized to sham vs. active in a 1:1 ratio. The second train of iTBS is active for all participants. After both iTBS trains are completed, repeat TMS-based measures, stop signal task and EEG data will be collected again. Visit 3 will be one week after visit 2. Visit 3 is a virtual computer-based visit to assess for any potential side effects.

ELIGIBILITY:
Inclusion Criteria:

1. ADHD diagnosis
2. Ages 12-17 years
3. Stimulant use is allowed but must be discontinued 24 hours prior to and during days of TMS visit

Exclusion Criteria:

1. Medical conditions contraindicated or associated with altered TMS risk profile, including history of intracranial pathology, epilepsy or seizure disorders, traumatic brain injury, brain tumor, stroke, intellectual disability, cerebral palsy, neurodegenerative conditions, hearing impairment, metallic objects in the head or any other serious medical condition
2. Presence of any implanted medical devices (e.g., ports, shunts, stimulators, cochlear implants)
3. For biological females who are post-menarche, current pregnancy based on urine pregnancy test.
4. Baseline problem of hearing impairment or chronic tinnitus
5. Any clinically significant finding on brain MRI
6. History of DSM-5 conduct disorder, major depressive disorder, bipolar disorder, obsessive compulsive disorder, anxiety disorder, psychotic disorder
7. Non-stimulant medication(s) for ADHD (e.g., alpha2 adrenergic agonist, atomoxetine, tricyclics)
8. Neuroleptic/antipsychotic medication(s)
9. Inability to undergo MRI
10. Active suicidality, history of suicidality, or high risk for suicide as assessed by a study physician
11. Substance abuse or dependence within the past year, based on 1) separate screening process of asking parent/guardian and participant, and 2) positive urine drug screen. Exception will be made for positive urine drug screen due to prescribed ADHD medication

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
TMS-based Short-Interval Intracortical Inhibition (SICI) | Immediately after each iTBS train
  This is a measure of primary motor cortex inhibitory activity.
EEG-based beta activity | Immediately after each iTBS train
  This is a measure of beta-band activity during performance of stop signal task.
TMS-based Cortical Silent Period (cSP) | Immediately after each iTBS train
  This is a measure of primary motor cortex inhibitory activity.
EEG-based alpha activity | Immediately after each iTBS train
  This is a measure of alpha-band activity during performance of stop signal task.

SECONDARY OUTCOMES:
Stop Signal Reaction Time | Immediately after each iTBS train
  This is a measure calculated from the stop signal task. This is an experimental measure of how well the participant can inhibit a motor action.

CONTACTS AND LOCATIONS:
Overall Officials: Steve W Wu, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No